CLINICAL TRIAL: NCT03235024
Title: A Prospective, Vehicle Controlled, Double Blind, Multicenter, Randomized, Phase II Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Subjects With Mild to Moderate Atopic Dermatitis
Brief Title: Study to Determine Safety and Efficacy of B244 in Subjects With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AOBiome LLC (Industry)
Collaborators: Veristat, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADB244-001
Record Dates: First submitted 2017-07-20; First posted 2017-08-01 (Actual); Results first posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Atopic Dermatitis Eczema

STUDY DESIGN:
Intervention Model Description: Randomization will be 1:1 so that equal number of patients will be treated in each Arm of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double blind study. Participants will be assigned to study treatment in accordance with the randomization schedule generated for the allocation of vehicle or B244 prior to the initiation of the trial. Randomization will be centrally-based and performed using an appropriate IWRS (an automated randomization system).
  Each participant scheduled to receive investigational product (IP) will receive a randomization number at the time of randomization. The randomization number will be used to identify the study medication kit assigned to the participant and indicate the treatment to be administered to that participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- B244 (Active Comparator): B244 suspension in 30ml/bottle
  Subjects will apply a total of 8 pumps of IP per application to all affected areas twice-a-day.
  Interventions: Biological: B244
- Vehicle (Placebo Comparator): Vehicle, 30ml/bottle
  Subjects will apply a total of 8 pumps of IP per application to all affected areas twice-a-day.
  Interventions: Biological: Vehicle

INTERVENTIONS:
Biological: B244 — B244 suspension
  Arms: B244
Biological: Vehicle — Vehicle suspension
  Arms: Vehicle

SUMMARY:
This is a Prospective, Vehicle Controlled, Double Blind, Multicenter, Randomized Phase II trial, comparing the effect of twice daily B244 application for 28 days vs vehicle application on treatment of mild to moderate AD

DETAILED DESCRIPTION:
This is a Prospective, Vehicle Controlled, Double Blind, Multicenter, Randomized Phase II trial, comparing the effect of twice daily B244 application for 28 days vs vehicle application on treatment of mild to moderate AD

At Screening and Baseline, all subjects must have atopic dermatitis, as defined by the Hanifin and Rajka criteria, which involves a minimum of 10% and a maximum of 30% body surface area, EASI score of 10 to 21 and pruritus visual analogue scale scores of ≥ 5 points on the VAS scale (at least moderate).

The total duration of the study will be approximately 9 weeks. Participants will report for a Screening visit and if all inclusion criteria are met, subjects will go through a two week washout phase before reporting for a Baseline visit.

Subjects will come in for visits at Day 14 (Week 2), Day 28 (Week 4). A final visit will be conducted at Day 42 (Week 6).

Efficacy will be assessed using Atopic Dermatitis Area and Severity Index (EASI) and Visual Analog Scale (VAS).

Blood and urine samples will be collected for standard safety laboratory tests and effect of the drug on inflammatory biomarkers. Participant's safety will be monitored throughout the study.

Investigators plan to enroll approximately 130 total patients.

Randomization will be 1:1 so that equal number of patients will be treated in each Arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥18 years of age
* In good general health as determined by a thorough medical history and physical examination, and vital signs
* Clinical diagnosis of mild to moderate atopic dermatitis according to the criteria of Hanifin and Rajka
* Mild to moderate Atopic Dermatitis area and severity index [EASI] 10-21
* A score of at least ≥ 5 points (moderate pruritus) on the VAS for pruritus
* A minimum of 10% and not more than 30% of the subjects' BSA affected by atopic dermatitis (affected is defined by physical examination findings: erythema, edema, scaling, lichenification, excoriation, with the excoriation serving as the physical examination correlate of pruritus)
* An IGA score of 2-3
* Patient has a history of AD for ≥12 months
* Ability to read and understand English and to provide written informed consent and authorization for protected health information disclosure

Exclusion Criteria:

* Pregnant and lactating women by urine pregnancy testing
* Subjects with any significant clinical abnormalities which may interfere with study participation
* Any skin condition which may interfere with evaluation of AD
* Atopic dermatitis only on the head or scalp
* Subjects with Atopic dermatitis on the face
* Unstable or actively infected atopic dermatitis
* Patients suffering from pruritus from conditions other than AD
* Patients with chronic pruritus due to systemic disease
* Patients with conditions requiring inhaled steroids
* Have concurrent skin disease of such severity in the study area that it could interfere with the study evaluation
* Have active skin infections on the treatment area
* Have received or planning to receive topical corticosteroids, topical coal tar, topical sulfur, topical PDE-4 inhibitors, topical antihistamines, topical antiseptics or antibiotics, topical antifungals, bleach baths, UVA or UVB phototherapy, oral/IV/inhaled steroids, antibiotics/antiviral/antifungal agents, oral probiotics, glucocorticoids treatment, calcineurin inhibitors, immunomodulating biologic agents, systemic glucocorticoids, systemic immunosuppressive or immunomodulatory agents within 2 weeks of Baseline visit.
* Current or recent history (≤3 months of systemic use of Otrexup™, Rasuvo®, Rheumatrex® and Trexall™ or its generic versions such as Methotrexate
* History of being seropositive for human immunodeficiency virus (HIV) at screening by laboratory testing at Screening
* History of being positive for Hepatitis B virus surface antigen (HBsAg) or positive Hepatitis C virus antibody (HCV Ab) at screening by laboratory testing at Screening
* History of renal disease
* Use of any investigational drugs within the previous 30 days prior to dosing or within a period of less than five times the drug's half-life, whichever is longer
* Use of any biologic within a period of 5 times its half-life
* Use of vinegar or bleach baths within 2 weeks of starting the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Ng-Cashin, MD, Study Director — Chief Medical Officer; Spiros Jamas, ScD, Study Director — AOBiome LLC
Locations (17):
- United States (17):
  - Central Research Associates, Birmingham, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Encino Research Center, Encino, California
  - Orange County Research Center, Tustin, California
  - Neostart Corporation d.b.a AGA Clinical Trials, Hialeah, Florida
  - Clinical Neuroscience Solution, Inc, Jacksonville, Florida
  - FXM Research Corp., Miami, Florida
  - FXM Research Miramar, Miramar, Florida
  - Clinical Neuroscience Solution, Inc, Orlando, Florida
  - Clinical Research Trials of Florida, Inc., Tampa, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - DeNova Research dba Arano, LLC, Chicago, Illinois
  - Clarkston Skin Research, Clarkston, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - LoveLace Scientific Resources, Albuquerque, New Mexico
  - Central Sooner Research, Norman, Oklahoma
  - Paddington Testing Co., Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- B244: B244 suspension (4x10E9 cells/ml) in 30ml/bottle
  Subjects will apply a total of 8 pumps of IP per application to all affected areas twice-a-day
  B244: B244 suspension
- Vehicle: Vehicle, 30ml/bottle
  Subjects will apply a total of 8 pumps of IP per application to all affected areas twice-a-day
  Vehicle: Vehicle suspension
Period: Overall Study
Arm/Group | B244 | Vehicle
Started | 61 | 61
Completed | 55 | 51
Not Completed | 6 | 10
Not completed — Adverse Event | 2 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population included all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | B244 | Vehicle | Total
Number analyzed (Participants) | 61 | 61 | 122
Age, Customized [Count of Participants; unit: Participants]
  < 30 years | 12 | 12 | 24
  ≥ 30 years | 49 | 49 | 98
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 44 | 80
  Male | 25 | 17 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 10 | 25
  Not Hispanic or Latino | 46 | 50 | 96
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 25 | 28 | 53
  White | 27 | 27 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Weight [Mean (Standard Deviation); unit: kg] | 85.420 (24.9020) | 85.542 (22.8794) | 85.481 (23.8132)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.027 (9.2237) | 30.551 (7.0286) | 30.289 (8.1702)
BMI Category [Count of Participants; unit: Participants]
  <20 kg/m^2 | 5 | 2 | 7
  20 to <25 kg/m^2 | 15 | 12 | 27
  25 to <30 kg/m^2 | 12 | 22 | 34
  ≥30 kg/m^2 | 29 | 25 | 54
Smoking History [Count of Participants; unit: Participants]
  Never | 32 | 39 | 71
  Former | 10 | 3 | 13
  Current | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Safety and tolerability endpoints will consist of all adverse events reporting during the study duration.
Time Frame: Baseline to Day 42
Population: Intent to Treat (ITT) population included all randomized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 61 | 61
Participants
  At Least 1 Treatment-Related TEAE | 2 | 4
  At Least 1 Treatment-Related Grade 3 or 4 TEAE | 0 | 0
  At Least 1 Treatment-Related Serious TEAE | 0 | 0

2. Secondary Outcome: Change in Eczema Area Severity Index (EASI) Score Between the Active and Vehicle Groups
Description: EASI is a validated tool used to measure the severity and extent of atopic dermatitis where clinical investigators assess the presence and severity of erythema, edema/papulation, excoriation, and lichenification (score 0-3: none=0, mild=1, moderate=2, severe=3, half-points allowed) and area of involvement (score 0-6: 0=0% involvement, 1=1-9% involvement, 2=10-29% involvement, 3=30-49% involvement, 4=50-69% involvement, 5=70-89% involvement, 6=90-100% involvement) across head and neck, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks). The EASI score can range from 0.0to 72.0 with increments of 0.1 and higher scores representing a greater severity of atopic dermatitis.
Time Frame: Baseline to Day 28
Population: Subjects from the Intent to Treat (ITT) population (all randomized subjects) that remained in the study at Day 28.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 56 | 51
score on a scale | -5.7 (4.46) | -5.9 (5.90)

3. Other Pre Specified Outcome: Change in Visual Analog Scale (VAS) Score for Pruritus Between the Active and Vehicle Group
Description: VAS (Visual Analog Scale) was performed as a measure of pruritus. The VAS is composed of a 10-cm line divided into a scale from 0 to 10, and subjects were to indicate the score that best represented the intensity of their itching over the 24-hour period before each visit where a higher score indicated greater severity in pruritus.
Time Frame: Baseline to Day 28
Population: Subjects from the Intent to Treat (ITT) population (all randomized subjects) that remained in the study at Day 28.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 56 | 51
score on a scale
  Week 2 Change from Baseline | -1.5 (2.23) | -0.6 (1.92)
  Week 4 Change from Baseline | -1.8 (2.81) | -1.4 (2.32)
Statistical Analysis 1: Comparison: B244 vs Vehicle; Test type: Equivalence — A sample size of 52 per group would achieve >80% power to reject the null hypothesis of equal means when the population mean difference is μ1 - μ2 = (-1.4) - (-5.3) = 3.9 with a standard deviation for both groups of 7.0 and with a significance level (alpha) of 0.025 using a 1-sided 2-sample equal variance t-test; p = 0.0228, t-test, 1 sided — At Week 2

4. Other Pre Specified Outcome: Change in the Skindex 16 Score Between the Active and Vehicle Group
Description: The Skindex 16 questionnaire was assigned to subjects to examine the relationship between the subject's skin health and quality of life. Subjects scored 16 questions from 0 to 6 (0=never bothered, 6=always bothered). Total scores could range between 0 to 96, where a higher score is associated with a worse quality of life.
Time Frame: Baseline to Day 28
Population: Subjects from the Intent to Treat (ITT) population (all randomized subjects) that remained in the study at Day 28.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 56 | 51
score on a scale | -0.2 (5.74) | -0.8 (1.28)

5. Other Pre Specified Outcome: Change in the IGA Score Between the Active and Vehicle Groups
Description: IGA (Investigator's Global Assessment) was used to assess the overall diseases severity on a scale of 0 to 4 (0=clear, 1=almost clear, 2=mild disease, 3=moderate disease, and 4=severe disease).
Time Frame: Baseline to Day 28
Population: Subjects from the Intent to Treat (ITT) population (all randomized subjects) that remained in the study at Day 28.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 56 | 51
score on a scale | -0.6 (0.82) | -0.7 (0.94)

6. Other Pre Specified Outcome: Difference in Actigraphy Scratching Event Count Per Hour During the Night Between the Active and Vehicle Group
Description: Subjects were provided two Actigraphy watches (one on each wrist) to accurately monitor subject's sleep, activity, and itching patterns.
Time Frame: Baseline to Day 28
Population: Subjects from the Intent to Treat (ITT) population (all randomized subjects) that remained in the study at Day 28 with data collected from Actigraphy watches (subjects with missing data were excluded from analysis).
Measure: Mean (Standard Deviation); unit: average scratching events per hour
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 7 | 4
average scratching events per hour | -3.4 (8.26) | 3 (7.92)

7. Other Pre Specified Outcome: Difference in Biomarkers Between Active and Vehicle Groups.
Description: To evaluate if B244 administration on the skin twice daily for 28 days will affect the levels of immune biomarkers.
Time Frame: Baseline and Day 28
Population: Data was not collected for this exploratory endpoint.
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Microbial Content
Description: Evaluate if B244 administration on skin twice daily will affect the microbial content on collected skin swab samples.
Time Frame: Baseline and Day 28
Population: Data was not collected for this exploratory endpoint.
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Week 6.
Description: All AEs occurring after signing of the ICF through study completion/early termination were to be reported. All AEs were to be recorded irrespective of whether they were considered drug related. AEs were to be evaluated by the Investigator at each visit for duration, intensity, and whether the event could have been associated with the IP or other causes. Adverse events believed to be possibly related to IP must have been followed until their resolution.
Arm/Group | B244 | Vehicle
All-Cause Mortality (participants affected / at risk) | 1/61 | 0/61
Serious Adverse Events (participants affected / at risk) | 1/61 | 0/61
Other Adverse Events (participants affected / at risk) | 16/61 | 14/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B244 (N=61) | Vehicle (N=61)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B244 (N=61) | Vehicle (N=61)
Bronchitis (Infections and infestations) | 2 | 0
Superinfection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Burning Sensation (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 3
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Lip Swelling (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Application site pain (General disorders) | 1 | 1
Application site pruritus (General disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Ear swelling (Ear and labyrinth disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Haemeoglobin decreased (Investigations) | 1 | 0
Uterine cyst (Reproductive system and breast disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall have 45 days to review the papers. Sponsor shall have the right to require Institution/Principal Investigator, as applicable, to remove specifically identified confidential information and/or delay the proposed publication or presentation for an additional one hundred twenty (120) days to enable Sponsor to seek patent protections.

DOCUMENTS (2):
  • Study Protocol (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/24/NCT03235024/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT03235024/SAP_001.pdf